CLINICAL TRIAL: NCT01449227
Title: Natural Course of Adhesive Capsulitis of Hip
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Joon Yoo, associate professor, Seoul National University Hospital
Other Study IDs: 1108-095-374
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis; hip
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this prospective study is to see the natural course of adhesive capsulitis of hip. The study is based on the hypothesis that the natural course of adhesive capsulitis of hip is similar to that of adhesive capsulitis of shoulder. This study is also based on a hypothesis that hip joint capsule stretching exercise will result in pain relief, recovery of hip range of motion in months.

ELIGIBILITY:
Inclusion Criteria:

* Painful hip with Limited range of motion (especially external rotation and abduction)

Exclusion Criteria:

* Acute trauma history
* hematologic abnormality (Rheumatologic disease, Autoimmune disease)
* Radiologic abnormality (joint degenerative change, calcification, loosebody, evidence of Femoroacetabular impingement, osteonecrosis of femoral head, etc)
* MRI: Extra-articular pathology

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample painful hip with limited ranage of motion
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-09

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea